CLINICAL TRIAL: NCT01144455
Title: A Randomized Cross-over Phase 2 Study of the Safety and Efficacy of Two Dose Levels of TH-302 in Combination With Gemcitabine Compared With Gemcitabine Alone in Previously Untreated Patients With Locally Advanced Unresectable or Metastatic Pancreatic Adenocarcinoma
Brief Title: Study of the Safety and Efficacy of TH-302 in Combination With Gemcitabine Compared With Gemcitabine Alone in Previously Untreated Patients With Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunoGenesis (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-404
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Locally Advanced Unresectable Pancreatic Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Locally Advanced Unresectable or Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gemcitabine (Active Comparator): Gemcitabine: 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle
  Interventions: Drug: Gemzar (Gemcitabine)
- 240 mg/m2 TH-302 + Gemcitabine (Experimental): TH-302: 240 mg/m2 administered IV over 30 minutes Day 1, 8, and 15 of each 28-day cycle
  Gemcitabine: 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle
  Interventions: Drug: Gemzar (Gemcitabine); Drug: TH-302
- 340 mg/m2 TH-302 + Gemcitabine (Experimental): TH-302: 340 mg/m2 of TH-302 be administered IV over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
  Gemcitabine: 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle
  Interventions: Drug: Gemzar (Gemcitabine); Drug: TH-302

INTERVENTIONS:
Drug: Gemzar (Gemcitabine) — 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle.
  Other Names: Gemcitabine
Drug: TH-302 — 240 mg/m2 of TH-302 will be administered IV over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
  Other Names: HAP; hypoxia activated prodrug
  Arms: 240 mg/m2 TH-302 + Gemcitabine
Drug: TH-302 — 340 mg/m2 of TH-302 will be administered IV over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
  Other Names: HAP; hypoxia activated prodrug
  Arms: 340 mg/m2 TH-302 + Gemcitabine

SUMMARY:
The purpose of this study is to determine whether Gemcitabine versus Gemcitabine and TH-302 are effective in the treatment of subjects with first-line metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
A hypoxic microenvironment is a characteristic of many solid tumors including pancreatic cancer. The presence of hypoxia in solid tumors is associated with a more malignant phenotype and resistance to chemotherapy. The hypoxia-activated prodrug, TH-302, is designed to selectively physiologically target the hypoxic microenvironment. There is an absence of therapeutic options for subjects with metastatic pancreatic cancer. Gemcitabine provides clinical benefit as a single agent, but median survival is about 6 months. Combining gemcitabine with TH-302 may enable the targeting of both the normoxic and hypoxic regions of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
3. Locally advanced unresectable or metastatic pancreatic ductal adenocarcinoma proven either by histology or cytology previously untreated with chemotherapy or systemic therapy other than:

   * Radiosensitizing doses of 5-fluorouracil;
   * Radiosensitizing doses of gemcitabine if relapse occurred at least 6 months after completion of gemcitabine;
   * Neoadjuvant chemotherapy if relapse occurred at least 6 months after surgical resection;
   * Adjuvant chemotherapy if relapse occurred at least 6 months after completion of adjuvant chemotherapy.
4. Measurable disease by RECIST 1.1 criteria (at least one target lesion outside of previous radiation fields)
5. Documentation of disease progression since any prior therapy
6. ECOG performance status of 0 or 1
7. Life expectancy of at least 3 months
8. Acceptable liver function:

   1. Bilirubin less than or equal to 1.5 times upper limit of normal
   2. AST (SGOT) and ALT (SGPT) less than or equal to 2.5 times upper limit of normal (ULN); if liver metastases are present, then less than or equal to 5 times ULN is allowed
9. Acceptable renal function:

   a. Serum creatinine less than or equal to ULN
10. Acceptable hematologic status (without hematologic support):

    1. ANC greater than or equal to 1500 cells/μL
    2. Platelet count greater than or equal to 100,000/μL
    3. Hemoglobin greater than or equal to 9.0 g/dL
11. All women of childbearing potential must have a negative serum pregnancy test and male and female subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose

Exclusion Criteria:

1. New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 6 months prior to Day 1, unstable arrhythmia or symptomatic peripheral arterial vascular disease
2. Known brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 3 months)
3. Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
4. Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause systemic or regional hypoxemia
5. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
6. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
7. Treatment of pancreatic cancer with radiation therapy or surgery within 4 weeks prior to study entry
8. Prior therapy with an hypoxic cytotoxin
9. Subjects who participated in an investigational drug or device study within 28 days prior to study entry
10. Known active infection with HIV, hepatitis B, or hepatitis
11. Subjects who have exhibited allergic reactions to a structural compound, biological agent, or formulation (containing solutol and/or propylene glycol) similar to TH- 302
12. Females who are pregnant or breast-feeding
13. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
14. Unwillingness or inability to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Borad, MD, Principal Investigator — Mayo Clinic; Shantan Reddy, MD, Principal Investigator — Lousiana Health Sciences Center - Shreveport
Locations (59):
- United States (59):
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Saint Edward Mercy Medical Center, Fort Smith, Arkansas
  - Disney Family Cancer Center, Burbank, California
  - Scripps Clinical Research Services, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Palo Alto Medical Foundation, Mountain View, California
  - Los Palos Oncology and Hematology, Salinas, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Hematology Oncology Associates, PC, Stamford, Connecticut
  - Florida Cancer Institute - New Hope, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Martin Memorial Cancer Center, Stuart, Florida
  - Atlanta Cancer Care, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University Melvin and Bren Simon Cancer, Indianapolis, Indiana
  - Purchase Cancer Group, Paducah, Kentucky
  - Medical Oncology, Baton Rouge, Louisiana
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - LSU Health Sciences Center - Feist Weiller Cancer Center, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Virgina Piper Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hematology and Oncology Associates at BridgePoint, Tupelo, Mississippi
  - Missouri Cancer Associates, Columbia, Missouri
  - Montana Cancer Institute Foundation, Missoula, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Oncology Hematology, P.C., Hudson, New York
  - Cancer Care of Western North Carolina, PA, Asheville, North Carolina
  - Alamance Oncology Hematolgy Associates, Burlington, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Oncology Specialists, PA, Hickory, North Carolina
  - Emerywood Hematology and Oncology, High Point, North Carolina
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Kaiser Permanente Northwest Region Oncology Hematology, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Greater Philadelphia Cancer and Hematology Specialists, P.C., Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Institute for Translational Oncology Research (ITOR), Greenville, South Carolina
  - Vanderbilt University Medical Center, Div. of Medical Oncology, Nashville, Tennessee
  - Texas Oncology-Beaumont, Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Oncology- Fort Worth - 12th Avenue, Fort Worth, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology-Sherman, Sherman, Texas
  - Texas Oncology-Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - Fairfax Northern Virginia Hematology Oncology, PC, Fairfax, Virginia
  - Providence Everett Regional Medical Center, Cancer Research Dept., Everett, Washington
  - Columbia Basin Hematology and Oncology0, Kennewick, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Borad MJ, Reddy SG, Bahary N, Uronis HE, Sigal D, Cohn AL, Schelman WR, Stephenson J Jr, Chiorean EG, Rosen PJ, Ulrich B, Dragovich T, Del Prete SA, Rarick M, Eng C, Kroll S, Ryan DP. Randomized Phase II Trial of Gemcitabine Plus TH-302 Versus Gemcitabine in Patients With Advanced Pancreatic Cancer. J Clin Oncol. 2015 May 1;33(13):1475-81. doi: 10.1200/JCO.2014.55.7504. Epub 2014 Dec 15. PMID 25512461
- See also: Threshold Pharmaceuticals, Inc — http://www.thresholdpharm.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- 240 mg/m2 TH-302 + Gemcitabine: TH-302: 240 mg/m2 administered IV over 30 minutes Day 1, 8, and 15 of each 28-day cycle
  Gemcitabine: 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle
  Gemzar (Gemcitabine): 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle.
  TH-302: 240 mg/m2 of TH-302 will be administered IV over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
- 340 mg/m2 TH-302 + Gemcitabine: TH-302: 340 mg/m2 of TH-302 be administered IV over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
  Gemcitabine: 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle
  Gemzar (Gemcitabine): 1,000 mg/m2 administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle.
  TH-302: 340 mg/m2 of TH-302 will be administered IV over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
Period: Overall Study
Arm/Group | Gemcitabine | 240 mg/m2 TH-302 + Gemcitabine | 340 mg/m2 TH-302 + Gemcitabine
Started | 69 | 71 | 74
Completed | 19 | 29 | 38
Not Completed | 50 | 42 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine | 240 mg/m2 TH-302 + Gemcitabine | 340 mg/m2 TH-302 + Gemcitabine | Total
Number analyzed (Participants) | 69 | 71 | 74 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 43 | 36 | 107
  >=65 years | 41 | 28 | 38 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 32 | 88
  Male | 40 | 44 | 42 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 5 | 12
  White | 62 | 64 | 67 | 193
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gemcitabine | 240 mg/m2 TH-302 + Gemcitabine | 340 mg/m2 TH-302 + Gemcitabine
Number analyzed (Participants) | 69 | 71 | 74
days | 111 [101 to 148] | 169 [130 to 211] | 183 [149 to 223]

ADVERSE EVENTS:
Arm/Group | Gemcitabine | 240 mg/m2 TH-302 + Gemcitabine | 340 mg/m2 TH-302 + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 37/69 | 35/71 | 43/74
Other Adverse Events (participants affected / at risk) | 69/69 | 71/71 | 74/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine (N=69) | 240 mg/m2 TH-302 + Gemcitabine (N=71) | 340 mg/m2 TH-302 + Gemcitabine (N=74)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (5)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 3 (4) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 4 (4)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (2) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4)
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (5)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (4)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 6 (6)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (5)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (7)
Bile duct obstruction (Hepatobiliary disorders) | 4 (4) | 4 (5) | 3 (3)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 5 (6) | 2 (3) | 2 (3)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 3 (3) | 1 (2) | 2 (3)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 2 (3)
Stent malfunction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine (N=69) | 240 mg/m2 TH-302 + Gemcitabine (N=71) | 340 mg/m2 TH-302 + Gemcitabine (N=74)
Urinary tract infection (Infections and infestations) | 7 (8) | 6 (8) | 17 (24)
Anaemia (Blood and lymphatic system disorders) | 30 (34) | 36 (60) | 38 (67)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 10 (18) | 11 (23)
Neutropenia (Blood and lymphatic system disorders) | 15 (21) | 27 (69) | 32 (113)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (32) | 36 (104) | 43 (216)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 17 (20) | 25 (32)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 11 (12) | 12 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (14) | 10 (12) | 16 (19)
Insomnia (Psychiatric disorders) | 8 (8) | 12 (12) | 10 (10)
Dizziness (Nervous system disorders) | 10 (10) | 4 (4) | 8 (13)
Dysgeusia (Nervous system disorders) | 5 (5) | 5 (5) | 12 (14)
Headache (Nervous system disorders) | 7 (7) | 7 (8) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 11 (12) | 9 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 16 (17) | 12 (15)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 10 (10) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 11 (11) | 21 (22) | 20 (23)
Abdominal pain upper (Gastrointestinal disorders) | 8 (10) | 9 (10) | 6 (9)
Constipation (Gastrointestinal disorders) | 22 (25) | 23 (28) | 25 (32)
Diarrhoea (Gastrointestinal disorders) | 17 (23) | 20 (23) | 27 (34)
Nausea (Gastrointestinal disorders) | 27 (32) | 26 (36) | 31 (47)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 13 (15) | 27 (35)
Vomiting (Gastrointestinal disorders) | 19 (27) | 15 (24) | 26 (39)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8) | 12 (12)
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 (4) | 18 (24) | 17 (26)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (13) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 9 (9) | 17 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (7) | 9 (10)
Chills (General disorders) | 7 (7) | 8 (13) | 12 (17)
Fatigue (General disorders) | 29 (34) | 42 (49) | 40 (51)
Oedema peripheral (General disorders) | 28 (35) | 26 (33) | 31 (42)
Pyrexia (General disorders) | 16 (21) | 18 (28) | 18 (25)
Alanine aminotransferase increased (Investigations) | 7 (8) | 10 (12) | 7 (10)
Blood alkaline phosphatase increased (Investigations) | 4 (5) | 17 (18) | 8 (9)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 11 (16) | 6 (8)
Neutrophil count decreased (Investigations) | 12 (17) | 16 (32) | 17 (36)
Platelet count decreased (Investigations) | 10 (13) | 17 (37) | 14 (28)
Weight decreased (Investigations) | 9 (9) | 7 (7) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No